CLINICAL TRIAL: NCT07068711
Title: Monitoring the Nutritional Status of Head and Neck Cancer Patients During Radiotherapy
Brief Title: Nutritional Status of Head and Neck Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zehra Margot Celik, Principal Investigator, Marmara University
Other Study IDs: 24062025-68
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Radiotherapy; Nutritional Status
Keywords: head and neck cancer; radiotherapy; nutritional status; quality of life; adverse events
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and Neck Cancer Patients: Patients over 18 years of age receiving radiotherapy

SUMMARY:
This study aims to monitor the nutritional status of patients with head and neck cancer undergoing radiotherapy treatment. Throughout the treatment process, patients' body composition, handgrip strength, food intake, quality of life, and treatment-related side effects will be regularly assessed. Measurements will include physical parameters like body weight, height, and waist circumference, as well as blood test results and nutrition-related questionnaires. By closely tracking these changes, the study seeks to identify early signs of nutritional deterioration and support timely interventions. The goal is to better understand nutrition-related challenges during treatment and ultimately improve patients' quality of life.

DETAILED DESCRIPTION:
This research focuses on evaluating the nutritional status of patients with head and neck cancer who are undergoing radiotherapy at Marmara University Pendik Research and Training Hospital, Radiation Oncology Clinic. Head and neck cancers often impair essential functions such as chewing, swallowing, and taste due to both tumor location and treatment side effects. These complications can severely reduce oral intake, leading to weight loss and malnutrition-factors known to negatively affect treatment outcomes and quality of life.

The study is planned to take place between July 1, 2025, and December 31, 2025, with the possibility of extending data collection until March 2026 if necessary. A total of 57 patients aged 18 years and older, who meet specific inclusion criteria and voluntarily consent to participate, will be enrolled.

Throughout the radiotherapy process and one month following its completion, participants' nutritional status and related health parameters will be systematically monitored. The following data collection methods will be used:

Body composition will be assessed weekly using bioelectrical impedance analysis (BIA), a non-invasive method that provides data on body fat, lean body mass, and water content.

Anthropometric measurements such as weight, height, waist and hip circumference, and mid-upper arm circumference will be performed.

Handgrip strength, a widely used indicator of muscle function and nutritional risk, will be measured weekly with a standardized dynamometer.

Dietary intake will be evaluated using 24-hour food recall interviews.

Nutritional risk screening tools, including the Patient-Generated Subjective Global Assessment (PG-SGA) and NUTRISCORE, will be administered to assess malnutrition risk.

Blood biochemical markers, including albumin, prealbumin, total protein, and C-reactive protein (CRP), will be recorded from patient files to assess nutritional and inflammatory status.

Quality of life will be measured using the validated EORTC QLQ-H&N35 questionnaire, specifically designed for head and neck cancer patients.

Treatment-related side effects (e.g., mucositis, dry mouth, swallowing difficulty) will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE).

Physical activity levels will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF).

All data will be collected through direct face-to-face interviews, clinical assessments, and medical record reviews. No experimental intervention will be administered; patients will receive their standard medical treatment as prescribed.

The primary goal of this study is to identify how radiotherapy affects the nutritional status of head and neck cancer patients, and how these changes relate to quality of life and treatment tolerance. Findings from this study will support the development of targeted nutritional strategies to improve patient outcomes and well-being during cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Diagnosed with head and neck cancer
* Receiving radiotherapy at Marmara University Pendik Training and Research Hospital, Radiation Oncology Clinic
* Willing to participate and able to provide written informed consent
* Able to communicate and cooperate during assessments

Exclusion Criteria:

* Patients for whom BIA measurement is not possible (e.g., caffeine intake within the last 4 hours, alcohol use in the last 24 hours, intense physical activity in the last 24-48 hours, menstruation, presence of pacemaker or metal implants)
* Patients with communication barriers or cognitive impairments
* Amputees or individuals with severe upper extremity deformities
* Patients with neuromuscular disorders, hemiplegia, rheumatoid arthritis, or moderate/severe neurological or cognitive impairment
* Patients receiving parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients from a University Hospital in Istanbul / Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
PG-SGA Score | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Nutritional status will be evaluated using the Patient-Generated Subjective Global Assessment (PG-SGA), a validated tool for assessing nutritional risk in cancer patients. The total score ranges from 0 to ≥35, with higher scores indicating worse nutritional status and greater need for nutritional intervention. A PG-SGA score >9 indicates a critical need for intervention. Unit of Measure: PG-SGA total score
Body Composition - BIA | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Body composition will be assessed using bioelectrical impedance analysis (BIA), which provides the following measurements: body weight, body fat mass, fat-free mass, total body water, intracellular water, and extracellular water. All measurements will be reported in kilograms (kg).
  Note: Body Mass Index (BMI) will be calculated and reported separately as a distinct outcome measure in kg/m².
  Unit of Measure: kg
Quality of Life - EORTC QLQ-H&N35 | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Patient-reported quality of life will be assessed using the EORTC QLQ-H&N35 questionnaire, a validated instrument developed by the European Organisation for Research and Treatment of Cancer (EORTC) for patients with head and neck cancer. Scores range from 0 to 100. Higher scores indicate a higher level of symptoms or problems, and therefore represent worse quality of life for symptom-related scales (e.g., pain, swallowing, speech). Unit of Measure: QLQ-H&N35 scale score (0-100)
Handgrip Strength | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Muscle strength will be measured using a handgrip dynamometer; the average of three trials will be used. Unit of Measure: kg
Dietary Intake - 24-Hour Food Recall | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Daily food intake will be recorded using the 24-hour recall method and analyzed using nutrition software to evaluate energy and nutrient adequacy.
Mid-Upper Arm Circumference (MUAC) | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Measured using a flexible tape at the midpoint between the shoulder and elbow. Unit of Measure: cm
Body Mass Index (BMI) | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Calculated from measured weight and height using the formula kg/m². Unit of Measure: kg/m²

SECONDARY OUTCOMES:
Malnutrition Risk - NUTRISCORE | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Malnutrition risk will be assessed using the NUTRISCORE screening tool, which evaluates nutritional status in oncology patients based on multiple risk factors. The total score ranges from 0 to 9, with higher scores indicating greater risk of malnutrition. A score ≥5 indicates a significant risk of malnutrition and the need for nutritional intervention. Unit of Measure: NUTRISCORE score
Waist Circumference | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Measured at the midpoint between the lower margin of the last rib and the iliac crest. Unit of Measure: cm
Hip Circumference | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Hip circumference will be measured at the widest part of the hips using a flexible, non-stretchable measuring tape while the participant is standing upright. Unit of Measure: cm
Waist-to-Hip Ratio (WHR) | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Calculated by dividing waist circumference by hip circumference.
Serum Albumin | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Laboratory blood test result used to assess protein status. Unit of Measure: g/dL
Prealbumin | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Laboratory blood test used to assess short-term changes in protein status. Unit of Measure: g/dL
Total Protein | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Laboratory measure of total serum proteins. Unit of Measure: g/dL
C-Reactive Protein (CRP) | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Marker of inflammation measured via blood test. Unit of Measure: mg/L
Treatment-Related Side Effects - CTCAE v5.0 | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Side effects will be evaluated and graded using the Common Terminology Criteria for Adverse Events (CTCAE).
  Unit of Measure: CTCAE grade (1-5)
Physical Activity - IPAQ-SF | Weekly during radiotherapy and at follow-up visit (1 month after treatment)
  Physical activity will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The total score is expressed in MET-minutes/week, calculated by multiplying the duration and frequency of walking, moderate, and vigorous activity by established MET values.
  Scores range from 0 to over 10,000 MET-minutes/week, depending on the participant's activity level. Higher scores reflect greater levels of physical activity, indicating a more favorable outcome.
  As per standard IPAQ guidelines, total physical activity can be categorized as:
  * Low (<600 MET-min/week)
  * Moderate (600-3,000 MET-min/week)
  * High (>3,000 MET-min/week) Unit of Measure: MET-minutes/week

CONTACTS AND LOCATIONS:
Overall Officials: Beste M Atasoy, Prof. Dr., Study Director — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital Radiation Oncology Clinic, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.